CLINICAL TRIAL: NCT06382324
Title: The Psychological Impact of Mindfulness Intervention to Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301280B0
Record Dates: First submitted 2024-04-01; First posted 2024-04-24 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament (Acl) Reconstruction
Keywords: Mindfulness; Napping; ACL injury; Return-to-sport; Polysomnography
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Intervention method:
  * Mindfulness napping group: listening to a record of mindfulness meditation practice for 40 minutes.
  * Control group: listening to light music for 40 minutes.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor of polysomnography did not know the data belongs which group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arem (Experimental): The patient randomized in the intervention arm will listen to the records of body scan for 40 minutes with polysomnography evaluation
  Interventions: Behavioral: mindfulness practice of body scan
- control arm (Placebo Comparator): listening to light music for 40 minutes with polysomnography evaluation
  Interventions: Behavioral: listening to light music

INTERVENTIONS:
Behavioral: mindfulness practice of body scan — Mindfulness intervention is one kind of psychological intervention. The founder of Mindfulness-Based Stress Reduction (MBSR), Jon Kabat-Zinn, described mindfulness as "awareness that arises through paying attention, on purpose, in the present moment, non-judgmentally" (Kabat-Zinn, 2003). Moreover, these attitudes can be nurtured through various practices such as body scan, meditation, yoga, mindful eating, and mindful walking. Mindfulness practices are recognized for their ability to alleviate stress among athletes and enhance their recovery capabilities (Li et al., 2019). Mindfulness practice has been shown to enhance athletes' performance (Chen et al., 2018)、 improve sleep quality (Rusch et al., 2019)，which in turn promotes emotional stability and physical recovery.
  Arms: intervention arem
Behavioral: listening to light music — listening to light music asa control
  Arms: control arm

SUMMARY:
Anterior cruciate ligament (ACL) reconstruction surgery is a common procedure performed by orthopedic surgeons. Postoperatively, patients often experience pain, muscle tension, and concerns about their ability to return to sports. These factors influence the recovery and return to sports capabilities of ACL patients. According to research, only 64% of patients are able to recover to their pre-injury level after surgery, and the success rate for returning to competitive sports is only 56%. Psychological factors during the recovery process may explain this disparity. ACL injury is associated with anxiety, pain reaction, and emotional disorders, with fear of re-injury being the most common obstacle to returning to sports, accounting for 19%. A study by Lentz et al. (2015) also found no significant differences in pain assessments between individuals who were afraid of re-injury and those who were able to return to sports at six months and one year after surgery. This suggests that fear of pain may limit activity and increase the risk of unsuccessful return to sports.

Mindfulness intervention is a psychological approach that involves non-judgmental awareness and focus on moment to moment. Mindfulness practice is known to reduce stress in athletes, promote recovery, enhance athletic performance, and improve sleep quality. Good sleep quality contributes to emotional stability and physical recovery. Even short daytime naps can be beneficial for athletes. A review of 37 studies of moderate quality found that daytime napping can improve physical and cognitive performance, psychological state, and nighttime sleep.

Therefore, investigators hypothesize that integrating mindfulness practice into daytime napping may lead to improved spirit upon waking, reduce sleep inertia, and over time, potentially increase the rate of return to sports after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Within the first month after ACL reconstruction without mindfulness practice experience

Exclusion Criteria:

* below 18 years old, previous exposure to mindfulness intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) | 5 times in one month after ACL reconstruction
  Electroencephalogram (EEG) is used to monitors patient's brain activities
Electrooculography (EOG) | 5 times in one month after ACL reconstruction
  Electrooculography (EOG) is a technique for measuring the movements of the human eyes. This helps to determine when REM sleep occurs, of which rapid eye movements are characteristic, and also essentially aids in determining when sleep occurs.
Electromyography (EMG) | 5 times in one month after ACL reconstruction
  Electromyography (EMG) is for evaluating and recording the electrical activity produced by skeletal muscles, uses four electrodes to measure muscle tension in the body as well as to monitor for an excessive amount of leg movements during sleep. Which are placed on patient's chim, R.anterior tibialis and L.anterior tibialis.
ECG (Electrocardiography) | 5 times in one month after ACL reconstruction
  ECG (Electrocardiography) measure the electrical activity of the heart.
Nasal/Oral airflow | 5 times in one month after ACL reconstruction
  Nasal/Oral airflow measured using pressure transducers, and/or a thermocouple, fitted in or near the nostrils
Thermistor | 5 times in one month after ACL reconstruction
  Thermistors are composed of a material that changes electrical resistance when exposed to temperature changes. As with the thermocouple, the temperature changes are sampled under a patient's nose or in front of the mouth.
Chest and abdominal belt | 5 times in one month after ACL reconstruction
  Chest and abdominal belt measured in concert with nasal/oral airflow by the use of belts. These belts expand and contract upon breathing effort.
Oximetry | 5 times in one month after ACL reconstruction
  Oximetry determines changes in blood oxygen levels which fits over a fingertip.
Snoring | 5 times in one month after ACL reconstruction
  Snoring and other noises. recorded with a sound probe over the neck.

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale (KSS) | 5 times in one month after ACL reconstruction
  The Karolinska Sleepiness Scale (KSS) was developed by Akerstedt and Gillberg in 1990. This scale uses a 1 to 9 scoring system where participants rate their current level of sleepiness. A lower score indicates higher alertness, while a higher score signifies increased somnolence.
  The Karolinska Sleepiness Scale (KSS) was developed by Akerstedt and Gillberg in 1990. This scale uses a 1 to 9 scoring system where participants rate their current level of sleepiness. A lower score indicates higher alertness, while a higher score signifies increased somnolence.
Five Facet Mindfulness Questionnaire (FFMQ) | before and after five times in one month after ACL reconstruction, 6-month, 12-month follow-up
  The FFMQ is a widely used self-report measure designed to assess an individual's mindfulness abilities and practices. It evaluates mindfulness across five specific facets, each representing a distinct aspect of mindfulness. n Observing: This facet involves paying attention to both external stimuli and internal experiences, such as thoughts and sensations, without judgment. n Describing: Participants describe their experiences, emotions, and thoughts with words and labels. It reflects the ability to put experiences into words. n Acting with Awareness: This facet measures the degree to which individuals engage in their daily activities with full presence and attention, avoiding automatic or mindless behaviors. n Non-Judging of Inner Experience: Participants evaluate their thoughts and feelings with an open and non-judgmental attitude, without labeling them as good or bad. n Non-reactivity to Inner Experience: This facet assesses an individual's ability to let thoughts and emotions arise
State-Trait Anxiety Inventory (STAIS) | before and after five times in one month after ACL reconstruction, 6-month, 12-month follow-up
  The STAI refers to a psychological assessment tool used to measure anxiety in adults. It consists of two separate subscales: the State Anxiety (S-Anxiety) subscale and the Trait Anxiety (T-Anxiety) subscale. Here's an overview of each subscale's content. S-Anxiety Subscale evaluates a person's current, temporary feelings of anxiety, which can vary based on situational factors. It consists of 20 items that describe how individuals feel at the present moment. Respondents rate their agreement with statements like "I am tense" or "I am worried" on a 4-point scale, ranging from "Not at all" to "Very much so." Higher scores indicate higher levels of current anxiety.
Anterior Cruciate Ligament Return to Sport After Injury Scale (ACL-RSI) (Short Version) | before and after five times in one month after ACL reconstruction, 6-month, 12-month follow-up
  The ACL-RSI is presently utilized for predicting the likelihood of athletes not returning to sport. It includes a series of questions that inquire about an individual's emotions, thoughts, and concerns related to their return to sports. It assesses aspects such as fear of reinjury, confidence in the injured knee's stability, perceived psychological readiness, and perceived risk of returning to sports. Participants rate their responses with higher scores indicating greater confidence and readiness to return to sports. Webster and Feller validated the short form of ACL-RSI, demonstrating its strong internal consistency and reliability in predicting return-to-sport outcomes, which was comparable to the full version. They also confirmed the validity of the abbreviated ACL-RSI version, proposing that athletes achieving scores exceeding 60% at 6 months post-surgery were significantly inclined to return to sport within 12 months. Conversely, individuals scoring below 39 points were less like

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Keelung, Taiwan